CLINICAL TRIAL: NCT00164593
Title: Youth Empowerment Solutions for Peaceful Communities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-4530; U49CE000348 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Violence; Juvenile Delinquency; Social Problems; Social Control, Informal
Keywords: Youth Violence; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Youth Empowerment Solutions for Peaceful Communities — YES is a multi-faceted program that (1) engages 7th and 8th graders in a youth development program, (2) enhances neighborhood organizations' ability to include youth in their activities, and (3) connects the youth participants and adults in neighborhood organizations (e.g., crime watches, block groups, neighborhood associations) to carry out neighborhood improvement activities (e.g., community gardens, parks cleanup).

SUMMARY:
This project is an evaluation of an intervention to involve youth in creating community change for peace promotion and violence prevention. The intervention, Youth Empowerment Solutions for Peaceful Communities (YES), includes three components: youth empowerment activities, neighborhood organization development, and community development projects that involve youth and organizations working together.

Hypothesis 1: Efforts to engage youth in the community change process will enhance their attachment to their community, reduce their problem behaviors, and begin to change norms among their peers about community violence and interpersonal problem solving.

Hypothesis 2: Efforts to make community-based organizations more youth-friendly and engaging will assist them to be more effective in reaching their community enhancement goals and will expand youth involvement in their mission.

Hypothesis 3: Efforts to create more health-enhancing land use (e.g., beautification, community gardens, parks development) will improve social organization (e.g., social capital, social cohesion, and social support), and reduce the level of violent incidents and crime in the community.

DETAILED DESCRIPTION:
The program will focus on youth and neighborhood organizations in one middle-school attendance area. A nearby middle-school attendance area will serve as a comparison community. We will assess change in community norms, fear, social cohesion and social capital using an existing community survey of adults in the two neighborhoods. A similar survey will assess changes in youths' social norms, fears, perceptions of social cohesion and social capital, as well as their violent behavior and ethnic identity and pride. We will also compare the intervention and comparison neighborhoods on several community-level measures including police incident data, hospital injury reports, school suspension data, and ratings of neighborhood qualities (e.g., vacant lots, community gardens, social interaction).

The long-term goals of YES are to:

1. modify environmental conditions that contribute to youth violence;
2. promote social norms supportive of community participation and nonviolence;
3. increase perceptions of neighborhood safety among residents; and
4. reduce the incidence of youth violence perpetration and victimization.

ELIGIBILITY:
Inclusion Criteria:

* 7th and 8th graders in the intervention middle-school attendance area
* Neighborhood organizations with at least 10 members serving the intervention middle-school attendance area

Exclusion Criteria:

* Students who have been suspended or expelled during the intervention period
* Neighborhood organizations that serve areas in both the intervention and comparison areas.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1142 (Actual)
Dates: Start 2005-04; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Youth Violence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Zimmerman, PhD, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States